CLINICAL TRIAL: NCT02435589
Title: The Effects of a Systematic Pain Assessment Approach on Critically Ill Patients Outcomes: A Randomized Interventional Clinical Study
Brief Title: The Effects of a Systematic Pain Assessment Approach on Critically Ill Patients Outcomes in ICU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cyprus University of Technology (Other)
Collaborators: Nicosia General Hospital (Other)
Responsible Party: Principal Investigator, Evanthia Georgiou, PhD student, Cyprus University of Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EX 043 - EP2
Record Dates: First submitted 2015-04-22; First posted 2015-05-06 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Intervention:
  1. systematic pain assessment
  2. Notification of results of assessments to nurses and physicians. Pain Assessments will be done with the use of 2 different behavioral pain tools by independent assessors and the results of the assessments will be notified to the nurses and physicians and their respond will be observed and documented
  Interventions: Other: Systematic pain assessment; Other: Notification of results of assessments
- Control Group (Active Comparator): Intervention. Systematic pain assessments. Assessments of pain will be done by independent assessors but results will not be notified to nurses or physicians
  Interventions: Other: Systematic pain assessment

INTERVENTIONS:
Other: Systematic pain assessment — Systematic assessment of pain twice daily with the use of 2 different behavioral pain tools (Behavioral Pain Scale - BPS, and Critical Care Pain Observation Tool - C-POT) for non-communicative patients and Numerical Rating Scale (NRS) 1-10 for communicative patients.
Other: Notification of results of assessments — Pain assessments will be carried out by independent investigators who will notify the results to ICU nurses and physicians and observe and document their reaction
  Arms: Intervention group

SUMMARY:
The purpose of this study is to investigate the effectiveness of a systematic approach to pain assessment in the critically ill patients' outcome The investigators hypothesize that, patients who will undergo systematic pain assessment and they will have their results notified to physicians and nurses, will demonstrate favorable effects on pain intensity, more efficient use of sedatives and analgesics, duration of mechanical ventilation, length of ICU stay, mortality, adverse events and complications, in relation to patients who will receive standard care alone. Moreover it is expected that they will demonstrate altered levels of plasma neuropeptides and biochemical markers in peripheral blood.

DETAILED DESCRIPTION:
Appropriate pain management depends on the systematic and comprehensive assessment of pain. Inaccurate pain assessment and the resulting inadequate treatment of pain in critically ill adults can have significant physiological and psychological consequences.

The investigators will examine whether a systematic pain assessment approach can improve patients outcomes.

120 ICU patients will be randomized either to control or intervention group. The control group will receive standard care plus pain assessments but nurses and physicians will be blind of these results. The intervention group will receive standard care plus systematic pain assessment and the results will be notified to nurses and physicians.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* All patients with an estimated source of pain or due to immunological process as trauma, surgery, or due to general factors such as endotracheal intubation, interventional catheters

Exclusion Criteria:

* Length of stay in the ICU <24 hours
* The patient receives neuromuscular blockers,
* The patient has a disease or condition, such as Guillain-Barre, peripheral neuropathy, which modifies sensory transmission of painful stimuli
* The patient has a disease or condition which complicates the assessment of pain behavior, such as decerebration or vegetative state, agitation> 3 in the Richmond Agitation sedation Scale (RASS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-03; Primary Completion 2015-11 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
a) Level of pain (intensity, incidence of high levels of pain with a numerical pain scale NRS> 6, Behavioral pain scale (BPS) > 5 and Critical pain observation Tool (C-POT) >2 | morning between 9:00-11: hrs, and afternoon between 4:00-6:00 hrs) for ten continuous days
To investigate the effect of the systematic assessment of pain among patients groups - control and intervention as to:The total dose, frequency of administration and the type of analgesics and sedatives received | every 24 hrs for ten continuous days

SECONDARY OUTCOMES:
Effect of the systematic evaluation of pain among patients groups - control and intervention as to:The degree of sedation/agitation | morning between 9:00-11: hrs, and afternoon between 4:00-6:00 hrs) for ten continuous days
Effect of the systematic evaluation of pain among patients groups - control and intervention as to:The levels of biochemical marker, cortisol, in the serum | morning 1st day intervention (one sample), 3rd day intervention (second sample), 5th day intervention (third sample)
Effect of the systematic evaluation of pain among patients groups - control and intervention as to:The levels of biochemical marker corticotrophin hormone -ACTH in the serum | morning 1st day intervention (one sample), 3rd day intervention (second sample), 5th day intervention (third sample)
Effect of the systematic evaluation of pain among patients groups - control and intervention as to: The levels of biochemical marker, b-endorphin in the serum | morning 1st day intervention (one sample), 3rd day intervention (second sample), 5th day intervention (third sample)
Effect of the systematic evaluation of pain among patients groups - control and intervention as to: The levels of neuropeptide Y | morning 1st day intervention (one sample), 3rd day intervention (second sample), 5th day intervention (third sample)
Effect of the systematic evaluation of pain among patients groups - control and intervention as to: The levels of neuropeptide , substance P in the serum | morning 1st day intervention (one sample), 3rd day intervention (second sample), 5th day intervention (third sample)
To investigate the effect of the systematic assessment of pain among patients groups - control and intervention as to duration of mechanical ventilation | Day and time of initiation of mechanical ventilation till the day and time of end of mechanical ventilation, up to six months.
To investigate the effect of the systematic assessment of pain among patients groups - control and intervention as to length of stay in the ICU | From the day of admission to ICU till the day of discharge from ICU, up to six months
To investigate the effect of the systematic assessment of pain among patients groups - control and intervention as to the occurrence of adverse events | every 24 hrs for ten continuous days

CONTACTS AND LOCATIONS:
Overall Officials: Evanthia G Georgiou, PhD Cand, Principal Investigator — Cyprus University of Technology
Locations (1):
- Nicosia General Hospital, Nicosia, Cyprus